CLINICAL TRIAL: NCT00422773
Title: Open Labeled, Multicenter Phase I/II Study Evaluating the Dose Escalation/Safety of Cetuximab and Oxaliplatin/5-FU/FA/Irinotecan as First-Line Treatment of Metastatic Colorectal Cancer
Brief Title: Safety of Cetuximab and Oxaliplatin/5-FU/FA/Irinotecan in First-Line Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Gunnar Folprecht, University Hospital Dresden, Medical Department I
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-COFI-014
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: phase I/II; cetuximab; oxaliplatin; irinotecan; 5-FU; chemotherapy; dose escalation; safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

ARMS (1):
- Cetuximab+ FOLFOXIRI (Experimental): Cetuximab and Irinotecan, Oxaliplatin, 5FU and Folinic acid
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Dose level Infusion time (h) Dose level unit 1 2 3 4 Cetuximab 2.0 mg/m² 500 500 500 500 Irinotecan, before oxaliplatin 1.0 mg/m² 95 125 165 180 Oxaliplatin, with folinic acid 2.0 mg/m² 85 85 85 85 Folinic acid, with folinic acid 2.0 mg/m² 400 400 400 400 5-FU Infusion 46.0 mg/m² 3200 3200 3200 3200
  Other Names: Cetuximab (C225, Erbitux by Merck)

SUMMARY:
The purpose of this study is to assess a maximal tolerable dose and to assess the safety of a chemotherapy-combination of cetuximab, irinotecan, oxaliplatin and 5-fluorouracil (5-FU)/folinic acid (FA) as first-line treatment for metastatic colorectal cancer.

DETAILED DESCRIPTION:
Dose escalation:

The first three patients will receive chemotherapy at the dose level 1 for 6 weeks (first three cycles). The dose will be escalated for the next patients by one dose level if none of the three patients at a dose level experience a dose-limiting toxicity (DLT) during the first six weeks. If one of the three patients has a DLT, an additional three patients will be enrolled at this dose level and the dose will be escalated if no additional patients experience a DLT. Otherwise, the dose escalation will be stopped, and the last dose will be regarded as the maximum tolerated dose (MTD). An intra-individual dose escalation is not planned.

Expanded cohort:

The MTD cohort will be expanded to a total of 16 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-resectable, histologically confirmed, epithelial growth factor receptor(EGFR)-positive or negative colorectal cancer
* WHO Performance status 0 or 1
* Signed written informed consent
* ≥ 18 years of age
* Effective contraception for both male and female subjects if the risk of conception exists
* Adequate bone marrow function: neutrophil blood cell count (NBC) ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L, hemoglobin ≥ 5.96 mmol/L (10 g/dL)
* Adequate liver and renal function: bilirubin ≤ 1.5 x upper normal level (UNL) and not increasing more than 25% within the last 4 weeks; ASAT and ALAT ≤ 5 x UNL; serum creatinine ≤ 1.5 x UNL.

Exclusion Criteria:

* Previous exposure to epidermal growth factor receptor-targeting therapy
* Previous chemotherapy for colorectal cancer except for adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment or 5-FU in combination with radiotherapy for rectal cancer
* Radiotherapy or major abdominal or thoracic surgery within the last 4 weeks before inclusion.
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy.
* Investigational agents or participation in clinical trials within 30 days before start of the treatment in study.
* Clinically relevant coronary disease or myocardial infarction within 12 months before study entry.
* Peripheral neuropathy > CTC (Common Toxicity Criteria)grade I
* Inflammatory bowel disease
* Previous malignancy (except for colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
* History of severe psychiatric illness
* Drug or alcohol abuse
* Known hypersensitivity reaction to any of the components of study treatment
* Pregnancy (absence to be confirmed by b-hCG (pregnancy-) test) or lactation period
* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess a maximal tolerable dose and the safety of a chemotherapy-combination of cetuximab, irinotecan, oxaliplatin and 5-FU/folinic acid as first-line treatment for metastatic colorectal cancer

SECONDARY OUTCOMES:
To assess the treatment regarding the following: feasibility, toxicity, response rate, resection rate, progression free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Folprecht, Dr., Principal Investigator — University Hospital Dresden, Medical Department I
Locations (3):
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus, Medizinische Klinik, Dresden, Saxony
  - Westdeutsches Tumorzentrum, Universitaetsklinikum Essen, Essen
  - Universitaetsklinik Mannheim GmbH, III. Medizinische Klinik, Mannheim

REFERENCES:
- [Derived] Folprecht G, Hamann S, Schutte K, Trarbach T, Stoehlmacher-Williams J, Ehninger G. Dose escalating study of cetuximab and 5-FU/folinic acid (FA)/oxaliplatin/irinotecan (FOLFOXIRI) in first line therapy of patients with metastatic colorectal cancer. BMC Cancer. 2014 Jul 19;14:521. doi: 10.1186/1471-2407-14-521. PMID 25038824